CLINICAL TRIAL: NCT04800159
Title: Cannabis Effects on Antiretroviral Therapy Pharmacokinetics and Neurotoxicity
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Center for Medicinal Cannabis Research (Other)
Responsible Party: Principal Investigator, Scott Letendre, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DA050491
Record Dates: First submitted 2021-02-19; First posted 2021-03-16 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: HIV; Cannabis Use
MeSH Terms: interventions — nabiximols; Dronabinol

STUDY DESIGN:
Intervention Model Description: The interventional component of the project (Phase 2) will have a randomized cross-over design that randomly assigns the order of the administration of the three study products (placebo, cannabis with higher concentration of tetrahydrocannabinol (THC) and lower concentration of cannabidiol (CBD), or cannabis with higher CBD concentration and lower THC concentration). The cannabis administration phase of this study will compare the study products to: 1) ART concentrations in blood and CSF and 2) measures of uridine 5'-diphospho-glucuronosyltransferase (UGT) activity.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will randomly receive one of the study products at each visit. All participants will receive all three of the study products. Allocation assignment of visits will be assigned using a randomization string provided by the statistician. The allocation schedule will be kept in the pharmacy and concealed from all other study personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- THC Cannabis (Active Comparator): 11.86% THC/ 1.12% CBD
  Interventions: Drug: THC Cannabis
- CBD Cannabis (Active Comparator): 0.35% THC/ 11.27% CBD
  Interventions: Drug: CBD Cannabis
- Placebo (Placebo Comparator): ≤ 0.03% THC/ ≤ 0.05% CBD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC Cannabis — Vaporization of cannabis
  Other Names: Marijuana
  Arms: THC Cannabis
Drug: CBD Cannabis — Vaporization of cannabis
  Other Names: Marijuana
  Arms: CBD Cannabis
Drug: Placebo — Vaporization of placebo
  Other Names: Marijuana with < 0.01% of THC and CBD
  Arms: Placebo

SUMMARY:
This study will address whether cannabis affects antiretroviral therapy (ART) drug concentrations, mood, and thinking. The project will have two phases. Phase 1 is an observational study, in which 120 people will be assessed to evaluate the effects of chronic cannabis use on ART drug concentrations, mood, and thinking. In Phase 2, the study will administer cannabis (or placebo) to 40 people to examine its acute effects on ART drug concentrations.

DETAILED DESCRIPTION:
People with human immunodeficiency virus (HIV) commonly use cannabis but whether cannabis affects the antiretroviral therapy (ART) that treats HIV is not well known. Cannabis can inhibit the activity of enzymes that metabolize and eliminate ART drugs from the body, which could result in higher concentrations of ART drugs in the body. Cannabis may also affect the distribution of ART drugs into the brain, which could have both beneficial (e.g., better HIV control) and detrimental (e.g., toxicity) effects. The effects of cannabis may are likely influenced by factors like how much is used (e.g., light vs. heavy use) and the route of use (e.g., smoked vs. ingested). This study will address whether cannabis affects ART concentrations in blood and cerebrospinal fluid as well as mood, and thinking. The project will have two phases. Phase 1 is an observational study, in which 120 people will be assessed once to evaluate the effects of chronic cannabis use on ART drug concentrations, mood, and thinking. In Phase 2, the study will administer cannabis (or placebo) to 40 people to examine its acute effects on ART drug concentrations.

ELIGIBILITY:
Inclusion Criteria for Study Entry:

1. Age 18 or older;
2. Capacity to provide informed consent;
3. Presence of HIV infection by a standard diagnostic test;
4. On a stable ART regimen for at least 1 month and with a suppressed viral load by self-report;
5. Willing to abstain from cannabis for at least 24 hours prior to the Phase 1 assessment.
6. Willing to abstain from grapefruit juice consumption for 4 weeks prior to the Phase 1 assessment.

Exclusion Criteria for Study Entry:

1. Traumatic brain injury, including head injury with loss of consciousness for greater than 30 minutes or resulting in neurologic complications;
2. Dementia, including Alzheimer's disease;
3. History of stroke with residual neurologic sequelae;
4. History of seizure disorder with a seizure in the past year;
5. Severe psychiatric disorder (e.g., schizophrenia) that might make the person's participation in the study unsafe;
6. Substance or alcohol use disorder in the past 3 months;
7. Contraindications to lumbar puncture for those consenting to lumbar puncture (e.g., coagulopathy).

Additional Inclusion Criteria for participation in the cannabis administration visits (Phase 2-interventional):

1. Treatment with an integrase inhibitor (i.e. dolutegravir);
2. Use of cannabis in the past 10 years without a severe adverse reaction (e.g., disorientation, paranoia, or hallucinations). The two-year cutoff is to ensure exposure to modern cannabis, which is more likely to match the drug concentrations administered in this study;
3. Willing to refrain from driving or operating heavy machinery after the visit; and
4. Willing to abstain from cannabis for at least 48 hours prior to the cannabis administration visits.
5. Willing to abstain from grapefruit juice consumption for 4 weeks prior to cannabis administration and during the administration visits

Additional Exclusion Criteria for participation in the cannabis administration visits (Phase 2-interventional):

1. Younger than 21 years due to problems with the use of cannabis in children and adolescents;
2. a respiratory condition that would be exacerbated by inhaling vaporized cannabis (e.g., asthma or chronic obstructive pulmonary disease) or limited lung capacity that would prevent the individual from performing the Foltin puff procedure;
3. History of cardiovascular disease, including myocardial infarction;
4. Uncontrolled hypertension with systolic blood pressure greater than 160 mm Hg or a diastolic blood pressure greater than 100 mm Hg prior to study product administration;
5. Resting pulse greater than 100 beats per minute prior to study product administration;
6. Pregnancy as determined by a human chorionic gonadotropin urine test, women who are lactating, or unwillingness to prevent pregnancy during the cannabis administration portion of the study (using birth control in women of child-bearing age). Acceptable methods of birth control are: oral contraceptive pills, diaphragm, condom, progestin implant, intrauterine contraceptive device, sterilization, etc;
7. Active opportunistic infection or malignancy requiring treatment;
8. Unintentional loss of 10% or more of body weight during the previous 6 months;
9. CD4+ T-cell count less than 200 cells/µL;
10. Estimated glomerular filtration rate < 30 mL/minute, indicative of renal dysfunction;
11. Hepatic transaminases > 2 times the upper limit of normal;
12. Current severe depressive symptoms (BDI-II score ≥ 31) or suicidal ideation;
13. Known sensitivity to Acetaminophen (the probe for UGT activity);
14. Current use of substances that could have adverse interactions with Acetaminophen or cannabis (e.g., grapefruit juice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
1a i. Antiretroviral therapy (ART) drug concentration in blood | Cross-sectional; measured before ART ingestion
  This will be done separately for participants who use ART drugs that are predominantly metabolized by cytochrome P450 (CYP) or uridine 5'-diphospho-glucuronosyltransferase (UGT) (estimated N=60 in each).
1a ii. Cerebrospinal fluid (CSF)/plasma ratio of ART drug concentrations | Cross-sectional; measured before ART ingestion
  This will be done separately for CYP and UGT groups (estimated N=60 in each).
1a iii. Change in ART drug concentrations in blood | 2 hours; measured before ART ingestion and at 2 hours after the ART ingestion
  This will be done separately for CYP and UGT groups (estimated N=60 in each).
1a iv. Change in CSF/plasma ratio of ART drug concentrations | 2 hours; measured before ART ingestion and at 2 hours after the ART ingestion
  This will be done separately for CYP and UGT groups (estimated N=60 in each).
1b i. Effects of placebo, THC, and CBD on ART drug concentration | 5 hours
  The investigators will use a mixed effects model to assess effects of acute cannabis treatment (placebo, THC, or CBD: N=40) on the area under the time-drug concentration curve.
1b ii. Effects of placebo, THC and CBD on the CSF/plasma ratio of ART drug concentrations | 5 hours
  The investigators will use a mixed effects model to assess effects of acute cannabis treatment (placebo, THC, or CBD: N=40) on CSF/plasma ratio of ART drug concentrations
1b iii. Comparison between the effects of placebo and THC on ART pharmacokinetics and between the effects of placebo and CBD on ART pharmacokinetics | 3 to 30 days
  Comparison of the the area under the time-concentration curve of ART pharmacokinetics for placebo and THC and placebo and CBD (n=40). The effect size will be measured as the standardized difference in mean outcomes between any two groups (Cohen's d).
1b iv. Comparison between the effects of placebo and CBD on the CSF/plasma ratio of ART drug concentrations and between the effects of placebo and THC on the CSF/plasma ratio of ART drug concentrations | 3 to 30 days
  Comparison of the the CSF/plasma ratio of ART drug concentrations with placebo and CBD and with placebo and THC (n=40). The effect size will be measured as the standardized difference in mean outcomes between any two groups (Cohen's d).
2a. Effects of chronic cannabis use on the CSF/serum albumin ratio and P-glycoprotein (P-gp) expression. | 3 to 30 days
  Multivariate linear regression will be used to regress markers of blood-brain barrier integrity and P-gp on cannabis use (n = 120), then ART drug concentrations on blood-brain barrier integrity and P-gp separately for the UGT and CYP groups
2b. Examine the correlation between ART concentration in CSF and blood during placebo treatment compared to THC and CBD administration. | 3 to 30 days
  The investigators will use a mixed effects model to evaluate the effects of cannabis on the correlation between ART concentration in CSF and blood (n = 40).
2c. Effects of THC or CBD on uridine 5'-diphospho-glucuronosyltransferase (UGT) activity compared to placebo. | 3 to 30 days
  The investigators will use a mixed effects model to examine the effects of drug treatment on UGT metabolism (n = 40).
3a. i. Correlation between CD4+ T-cell count and ART drug concentration. | Up to 5 weeks: baseline to administration visits
  Multivariable linear regressions will be used for testing correlation between CD4+ T-cell count and ART drug concentration (N=60 in each UGT and CYP groups).
3a. ii. Correlation between HIV DNA and ART drug concentration. | Up to 5 weeks: baseline to administration visits
  Multivariable logistic regressions will be used for testing correlation between HIV DNA and ART drug concentration (N=60 in each UGT and CYP groups).
3b i. Effects of cannabis use on the correlation between ART and neurocognitive performance. | 3 to 30 days
  The total cognitive outcome from the National Institutes of Health Toolbox will be regressed in multivariable models on ART drug concentration and cannabis use, their interaction, and known confounders and relevant covariates. Values range from 0 to 100 with lower values being worse.
3b ii. Effects of cannabis use on the correlation between ART and depression. | 3 to 30 days
  Depression (measured with the Beck Depression Inventory-II) will be regressed in multivariable models on ART drug concentration and cannabis use, their interaction, and known confounders and relevant covariates.
3b iii. Effects of cannabis use on the correlation between ART and emotional health. | 3 to 30 days
  The National Institutes of Health Toolbox-Emotional Battery outcome, Negative Affect, will be regressed in multivariable models on ART drug concentration and cannabis use, their interaction, and known confounders and relevant covariates. This measure ranges between 0 and 100 with higher values reflecting more Negative Affect.
3b iv. Effects of cannabis use on the correlation between ART and emotional health. | 3 to 30 days
  The National Institutes of Health Toolbox-Emotional Battery outcome, Social Satisfaction, will be regressed in multivariable models on ART drug concentration and cannabis use, their interaction, and known confounders and relevant covariates. This measure ranges between 0 and 100 with lower values reflecting worse Social Satisfaction.
3b v. Effects of cannabis use on the correlation between ART and emotional health. | 3 to 30 days
  The National Institutes of Health Toolbox-Emotional Battery outcome, Psychological Wellbeing, will be regressed in multivariable models on ART drug concentration and cannabis use, their interaction, and known confounders and relevant covariates. This measure ranges between 0 and 100 with lower values reflecting worse Psychological Wellbeing.
3b vi. Effects of cannabis use on the correlation between ART and neurotoxicity. | 3 to 30 days
  A measure of neurotoxicity (mitochondrial DNA) will be regressed in multivariable models on ART drug concentration and cannabis use, their interaction, and known confounders and relevant covariates.
3b vii. Effects of cannabis use on the correlation between ART and neurotoxicity. | 3 to 30 days
  A measure of neurotoxicity (8-hydroxydeoxyguanosine) will be regressed in multivariable models on ART drug concentration and cannabis use, their interaction, and known confounders and relevant covariates.
3b viii. Effects of cannabis use on the correlation between ART and neurotoxicity. | 3 to 30 days
  A measure of neurotoxicity (F2-isoprostane) will be regressed in multivariable models on ART drug concentration and cannabis use, their interaction, and known confounders and relevant covariates.

SECONDARY OUTCOMES:
1b v. Comparison between the effects of THC and CBD on ART pharmacokinetics. | 3 to 30 days
  Comparison of the treatment arm to the the area under the time-concentration curve of ART pharmacokinetics (n=40).
1b vi. Comparison between the effects of THC and CBD on the CSF/plasma ratio of ART drug concentrations. | 3 to 30 days
  Comparison of treatment arm to the CSF/plasma ratio of ART drug concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Letendre, MD, Principal Investigator — UCSD
Locations (1):
- Ucsd Hnrp-Cmcr, San Diego, California, United States